CLINICAL TRIAL: NCT05500638
Title: Effect of Virtual Reality Based Seizure Management Education Program for Parents (VR-ESMEPP) on Seizure Management: Randomized Controlled Trial
Brief Title: Effect of VR-ESMEPP on Parents' Seizure Management
Acronym: VR-ESMEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ayşegül İşler Dalgıç, Prof., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012-KAEK-20-730
Record Dates: First submitted 2022-08-08; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Virtual Reality; Epilepsy; Seizure; Child; Nurse; Parents
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: A total of two groups as 1 intervention (virtual reality) and control group (usual care)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: At the end of the study, the data of the participants at T0, T1 and T2 times were recorded and stored by the system. The participants, the researcher and the instructor who made the statistics did not see the results of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Firstly, the intervention group was administered the pretest, then the training program (VR-ESMEPP), and a posttest immediately following the training. The participants were monitored on the 15th day.
  Interventions: Behavioral: Virtual Reality
- Control Group (No Intervention): For the control group, a pretest, routine outpatient clinical practices, and a posttest were carried out; and the participants were monitored on day 15. They took usual care.

INTERVENTIONS:
Behavioral: Virtual Reality — At this stage, trainings were given for epileptic seizures. Parents were asked to wear SG glasses and they were trained on the correct approach to seizures over the Focal to bilateral tonic-clonic seizure scenario integrated into the SG glasses. The clinic and process of focal to bilateral tonic-clonic seizure and the training of what to do and not to do during the seizure were given again through SG glasses. Parents interfered with the patient scenario many times during their free work time and had the chance to interfere with the seizure again and again by restarting the seizure.
  Arms: Virtual Reality Group

SUMMARY:
Objective: This study aims to evaluate the knowledge, skills, and motivation of parents regarding management of epileptic seizures, by developing a "Virtual Reality Based Seizure Management Education Program for Parents (VR-ESMEPP).

Method: This study is a double-blinded, pretest-posttest, observational randomized controlled study. The administration stage of the study was conducted between September 2018-February 2020 with parents of 91 children who were diagnosed with epilepsy and were being followed in the Pediatric Neurology Outpatient Department of Akdeniz University Hospital. The parents were distributed into groups with simple randomization (VR Group n=45-Control Group n=46). During the preparation stage of the study, data collection tools "Management-of-Epileptic Seizure-Training-Program-Prepared-with-Virtual-Reality-Technology" and "Patient Scenario Regarding Secondary Generalized Tonic-Clonic Epileptic Scenario with Aura" were prepared and integrated into the virtual reality glasses. In the administration stage, the intervention group was administered the pretest, then the training program, and a posttest immediately following the training. The participants were monitored on the 15th day. For the control group, a pretest, routine outpatient clinical practices, and a posttest were carried out; and the participants were monitored on day 15. In both groups, data were obtained with data collection tools that were integrated into the virtual reality glasses. An approval from the Ethics Committee of Akdeniz University, a written permission from the Akdeniz University Hospital, and informed consent from the parents were obtained to conduct the study.

DETAILED DESCRIPTION:
Objective: Parents of children with epilepsy need support when managing epileptic seizures outside medical-care-center-settings. Previously developed training programs only provide information-based support. Therefore, within the scope of the VR-ESMEPP, a conceptual framework was developed in this study with the aim of developing parents' skills and motivation as well as providing them information regarding seizure management.

Methods: The conceptual framework of the VR-ESMEPP was developed in four steps. In step 1, a scenario was developed wherein an epileptic pediatric patient is having a seizure. The selected seizure type was generalized-tonic-clonic-seizure, which is the most common and most skill-intensive type of tonic-clonic-seizure. In step 2, data collection tools related to epileptic seizure management were developed for parents. These tools included Child and Parent Introductory Form, Parental Information Assessment Form for Epileptic Seizure Management, and Parental Skills Assessment Form for Epileptic Seizure Management. In step 3, the conceptual framework and data collection tools developed were confirmed by a group of 10 specialists consisting of physicians and pediatric nurses working in the field of pediatric neurology. In step 4, the epileptic-pediatric-patient-scenario and data collection tools confirmed by experts were programmed into an application by a software company and integrated into virtual reality headsets.

ELIGIBILITY:
Inclusion Criteria:

* Parents who had a child with a diagnosis of "focal to bilateral tonic-clonic" seizure, who could speak Turkish, who had no limitations in hearing, vision and hand motor skills in order to use the virtual reality glasses effectively, were included in the study.

Exclusion Criteria:

* Participants outside of these criteria were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Effects on knowledge about epilepsy change | baseline, pre-intervention
  Parental Information Assessment Form for Epileptic Seizure Management. This form was prepared by researchers in line with the relevant literature to evaluate the parents' level of knowledge related to seizure intervention. The form consists of a total of 22 binary Likert-type questions answered as "True" or "False." Four questions included reverse statements.
Effects on knowledge about epilepsy change | immediately after the intervention
  Parental Information Assessment Form for Epileptic Seizure Management. This form was prepared by researchers in line with the relevant literature to evaluate the parents' level of knowledge related to seizure intervention. The form consists of a total of 22 binary Likert-type questions answered as "True" or "False." Four questions included reverse statements.
Effects on knowledge about epilepsy change | 15 days after the intervention
  Parental Information Assessment Form for Epileptic Seizure Management. This form was prepared by researchers in line with the relevant literature to evaluate the parents' level of knowledge related to seizure intervention. The form consists of a total of 22 binary Likert-type questions answered as "True" or "False." Four questions included reverse statements.
Effects on skill about epileptic seizure time | baseline, pre-intervention
  Parental Skills Assessment Form for Epileptic Seizure Management. This form consists of seven questions prepared by researchers in line with the relevant literature in order to evaluate the seizure intervention-related skills of parents. These seven questions focus on the seven skills that parents are expected to have to perform a seizure intervention. These skills include assessing the child's consciousness when the seizure begins, recording seizure time, removing close objects that may cause injury, loosening the child's clothes, turning the head sideways, and calling for emergency help (calling an ambulance). The expert opinions were obtained regarding the pediatric-patient-scenario and data collection tools developed by the researchers.
Effects on skill about epileptic seizure time | immediately after the intervention
  Parental Skills Assessment Form for Epileptic Seizure Management. This form consists of seven questions prepared by researchers in line with the relevant literature in order to evaluate the seizure intervention-related skills of parents. These seven questions focus on the seven skills that parents are expected to have to perform a seizure intervention. These skills include assessing the child's consciousness when the seizure begins, recording seizure time, removing close objects that may cause injury, loosening the child's clothes, turning the head sideways, and calling for emergency help (calling an ambulance). The expert opinions were obtained regarding the pediatric-patient-scenario and data collection tools developed by the researchers.
Effects on skill about epileptic seizure time | 15 days after the intervention
  Parental Skills Assessment Form for Epileptic Seizure Management. This form consists of seven questions prepared by researchers in line with the relevant literature in order to evaluate the seizure intervention-related skills of parents. These seven questions focus on the seven skills that parents are expected to have to perform a seizure intervention. These skills include assessing the child's consciousness when the seizure begins, recording seizure time, removing close objects that may cause injury, loosening the child's clothes, turning the head sideways, and calling for emergency help (calling an ambulance).

SECONDARY OUTCOMES:
Effects on motivation change | baseline, pre-intervention
  Instructional Materials Motivation Survey. for analog and digital learning environments. 5-point Likert Scale (1 (or A) = Not true; 2 (or B) = Slightly true; 3 (or C) = Moderately true; 4 (or D) = Mostly true; 5 (or E) = Very true). Attention: Cronbachs α: .83 Relevance: Cronbachs α: .81 Satisfaction: Cronbachs α: .92 Confidence: Cronbachs α: . 90
Effects on motivation change | immediately after the intervention
  Instructional Materials Motivation Survey. for analog and digital learning environments. 5-point Likert Scale (1 (or A) = Not true; 2 (or B) = Slightly true; 3 (or C) = Moderately true; 4 (or D) = Mostly true; 5 (or E) = Very true). Attention: Cronbachs α: .83 Relevance: Cronbachs α: .81 Satisfaction: Cronbachs α: .92 Confidence: Cronbachs α: . 90
Effects on motivation change | 15 days after the intervention
  Instructional Materials Motivation Survey. for analog and digital learning environments. 5-point Likert Scale (1 (or A) = Not true; 2 (or B) = Slightly true; 3 (or C) = Moderately true; 4. (or D) = Mostly true; 5 (or E) = Very true). Attention: Cronbachs α: .83 Relevance: Cronbachs α: .81 Satisfaction: Cronbachs α: .92 Confidence: Cronbachs α: . 90

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül İşler Dalgıç, Prof., Study Director — Akdeniz University
Locations (1):
- Aysegul ISLER DALGIC, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No